CLINICAL TRIAL: NCT01571687
Title: Pik Lenin High Altitude Research Expedition 2009, a Follow-up Project of the Muztagh Ata High Altitude Research Expedition 2005
Brief Title: Pik Lenin High Altitude Research Expedition 2009
Acronym: PLHARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Kantonsspital Aarau (Other); Lotteriefonds des Kantons Aarau (Unknown); Schweizer Gesellschaft für Gebirgsmedizin (Unknown); University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2008/071; 07.09.34 (Other: University Hospital Berne)
Record Dates: First submitted 2012-03-28; First posted 2012-04-05 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Oxidative Stress; Cell-derived Microparticles
Keywords: expedition; hypoxia; blood coagulation disorders; cell-derived microparticles; oxidative stress; N-Acetylcystein; vitamins
MeSH Terms: conditions — Hypoxia; Blood Coagulation Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- antioxidant supplements (Active Comparator): 800 I.E. Vitamin E, 1000mg Vitamin C, 200000 I.E. Vitamin A, 600mg Acetylcystein.
  Interventions: Dietary Supplement: antioxidant supplements
- Placebo (Placebo Comparator): identically appearing placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: antioxidant supplements — Intake of 6 tablets daily containing: 800 I.E. Vitamin E, 1000mg Vitamin C, 200000 I.E. Vitamin A, 600mg Acetylcystein.
  Arms: antioxidant supplements
Dietary Supplement: Placebo — Intake of 6 identically appearing tablets daily containing placebo
  Arms: Placebo

SUMMARY:
Exposure to hypobaric hypoxia demands maximum effort of the body and can lead to high altitude illnesses. Recently, there is rising interest on coagulation activation during trekking and mountaineering in higher regions and on development of oxidative stress due to hypoxia. 30 volunteers have been examined during an high altitude research expedition to the 7134m high mount Pik Lenin in Kyrgyzstan to investigate mechanisms of coagulation activation and effects of antioxidant supplements on oxidative stress.

DETAILED DESCRIPTION:
Reactions to acute exposure to high altitude and the process of acclimatization has been of scientific interest since many years. High altitude illnesses are specified by three different entities: acute mountain sickness (AMS), high altitude pulmonary edema (HAPE) and high altitude cerebral edema (HACE). Prevalence of AMS is known to be between 10 to 20% for altitudes between 4000 and 5000m, increasing significantly in higher altitude. The prevalence depends on the ascent rate, individual susceptibility and physical exhaustion.

Although mechanisms leading to high altitude illnesses are not yet completely clear some progress has been made. It is well accepted that excessive pulmonary hypertension may lead to HAPE. Furthermore, there is rising evidence about endothelial dysfunction being involved in disease progression. Some cellular and molecular mechanisms of acute (hypobaric) hypoxia, possibly leading to endothelial dysfunction, have been studied in a few experimental and field settings. Paradoxical increase in systemic oxidative stress is seen under hypoxic conditions, such as high altitude stay. Reactive oxygen species (ROS) could be demonstrated in many endothelial disorders and capillary leakage syndromes such as septicaemia, myocardial infarct and stroke. Furthermore, coagulation activation might result from endothelial dysfunction but also amplify endothelial interruption. Still, most of our knowledge concerning effects of hypoxia in general but also concerning oxidative stress is from in vitro studies (e.g. cancer cells).

In the context of a high altitude expedition human subjects can safely be submitted to prolonged hypoxia to explore generation of ROS and extent of procoagulatory state.

Objective

The purpose of our study is to confirm excessive oxidative stress found in our previous study in 2005 and to investigate whether oxidative stress during high altitude exposure can be modified by dietary supplementations of specific antioxidants. Moreover, we like to study mechanisms of coagulation activation by assessing extent of thrombocytic and endothelial microparticles.

Methods

After approval of the study by the regional ethics committee, written informed consent has been obtained from 30 healthy volunteers (low land residents with mountaineering experience, age 18-65 years). After baseline testing, double-blind randomization into 2 groups of 15 persons took place. One group received oral medication with vitamin E, vitamin C, vitamin A and acetylcystein daily, while the other group was provided with an identical appearing placebo preparation. Substitution started 2 month before the expedition. After examination at "ground 0" in Zurich (409m) all members underwent testing in Base Camp (3550m), twice in advanced Base Camp (4550m), in Camp 1 (5430m), and in Camp 2 (6265m). Beside blood sampling, clinical examinations were performed. Metabolomics, a mass-spectrometry based analysis, for measurement of oxidative stress, will be performed. In a subgroup microparticles will be detected by annexin V based ELISA and by flow cytometry using specific antibodies.

ELIGIBILITY:
Inclusion Criteria:

* good health status
* age 18-65
* mountaineering experience

Exclusion Criteria:

* any metabolic disorders
* regular drug intake
* any disease of the lungs
* any disease of the heart
* any renal abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in oxidative stress | during expedition, up to 22 days

SECONDARY OUTCOMES:
Change from baseline in coagulation activation | during expedition, up to 22 days
Change from baseline in acute mountain sickness score | during expedition, up to 22 days
Change from baseline in oxygen saturation in blood | during expedition, up to 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Andreas R Huber, Prof. Dr. med., Study Chair — Center of Laboratory Medicine Cantonal Hospital Aarau and University of Bern; Jacqueline Pichler Hefti, Dr. med., Principal Investigator — Division of Pneumology, Inselspital Bern, Universityhospital Bern
Locations (1):
- Center of Laboratory Medicine Cantonal Hospital Aarau and University of Bern, Aarau, Switzerland

REFERENCES:
- [Background] Basnyat B, Murdoch DR. High-altitude illness. Lancet. 2003 Jun 7;361(9373):1967-74. doi: 10.1016/S0140-6736(03)13591-X. PMID 12801752
- [Background] Hackett PH, Rennie D, Levine HD. The incidence, importance, and prophylaxis of acute mountain sickness. Lancet. 1976 Nov 27;2(7996):1149-55. doi: 10.1016/s0140-6736(76)91677-9. PMID 62991
- [Background] Taniyama Y, Griendling KK. Reactive oxygen species in the vasculature: molecular and cellular mechanisms. Hypertension. 2003 Dec;42(6):1075-81. doi: 10.1161/01.HYP.0000100443.09293.4F. Epub 2003 Oct 27. PMID 14581295
- [Background] Huet O, Dupic L, Harrois A, Duranteau J. Oxidative stress and endothelial dysfunction during sepsis. Front Biosci (Landmark Ed). 2011 Jan 1;16(5):1986-95. doi: 10.2741/3835. PMID 21196278
- [Result] Pichler Hefti J, Risch L, Hefti U, Scharrer I, Risch G, Merz TM, Turk A, Bosch MM, Barthelmess D, Schoch O, Maggiorini M, Huber AR. Changes of coagulation parameters during high altitude expedition. Swiss Med Wkly. 2010 Feb 20;140(7-8):111-7. doi: 10.4414/smw.2010.12910. PMID 19950043